CLINICAL TRIAL: NCT02426437
Title: How Does Early Rehabilitation Affect Patient-centred Health Outcomes and Cardiovascular Risk in COPD Patients
Brief Title: Examining Pulmonary Rehabilitation on Discharged COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00038838-2; AIHS-CRIO Project Grant (Other: Alberta Innovated Health Solutions (AIHS))
Record Dates: First submitted 2015-03-17; First posted 2015-04-27 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Acute Exacerbation of COPD (AECOPD); COPD; Emphysema; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Early Pulmonary Rehabilitation (EPR) (Other): Patients randomized to EPR will be enrolled into the Breath Easy pulmonary rehabilitation (PR) program at the Centre for Lung Health within 1 month of discharge. They will proceed through the program in a typical fashion.
  Interventions: Other: Pulmonary Rehabilitation (PR)
- Late Pulmonary Rehabilitation (LPR) (Other): Patients randomized to LPR will be enrolled into the Breath Easy pulmonary rehabilitation (PR) program at the Centre for Lung Health within 3 months of discharge. They will proceed through the program in a typical fashion.
  Interventions: Other: Pulmonary Rehabilitation (PR)
- Usual Care (Other): Usual care patients will be followed-up by their most responsible physician as determined by the admitting team.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Pulmonary Rehabilitation (PR) — Patients enrolled in PR will undergo a 6-8 week rehabilitation program.
  Arms: Early Pulmonary Rehabilitation (EPR); Late Pulmonary Rehabilitation (LPR)
Other: Usual Care — Patients enrolled in usual care will be followed-up by their most responsible physician as determined by the admitting team.
  Arms: Usual Care

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic lung disease primarily caused by smoking. COPD creates a tremendous burden to the healthcare system, as disease exacerbations result in frequent, prolonged hospitalizations. While originally considered a disease specific to the lung, data has shown that COPD is associated with substantial cardiovascular (CV) morbidity and mortality. Exacerbations of COPD requiring hospitalization result in marked patient deterioration, and heightened CV risk. The cause of the increased CV risk with stable COPD, and the exaggerated CV risk during exacerbations of the disease are unknown; however, it may be due to chronic inflammation which is exacerbated with a flare-up of the disease, and/or chronic inactivity which is similarly worsened with bed-rest during a hospitalization. Despite the impact of COPD on healthcare, there are relatively few studies examining how COPD inpatient care impacts on patient outcomes, inflammation and CV risk. Disease management programs, such as pulmonary rehabilitation and patient self-management education, are part of guideline therapy for COPD; however, these are not regularly implemented following a hospitalization, and how these interventions affect patient outcomes, behavior, physical activity, inflammation and CV risk have not been well studied. The proposed long-term project will examine how early referral to chronic disease management programs after hospital discharge, affect patient outcomes. This study will provide invaluable information about outpatient management for a disease which has a tremendous impact on healthcare.

DETAILED DESCRIPTION:
Purpose: To examine the impact of early pulmonary rehabilitation (PR) following hospital discharge on QoL, pulmonary/CV outcomes and AECOPD hospitalizations.

Rationale: In addition to typical improvements in QoL and exercise tolerance, studies have shown that PR increases self-efficacy and physical activity while reducing CV risk in stable COPD patients. Patients recently discharge from hospital following AECOPD represent the sickest patients with greatly reduced QoL, exercise tolerance, self-efficacy and physical activity. Exactly how these improve with PR following a hospitalization requires examination.

Hypothesis: Patients who receive early PR will have improved QoL, pulmonary/CV outcomes and less hospitalizations for COPD in the 6 months following hospital discharge. PR will improve self efficacy, physical activity and QoL while reducing CV risk as compared to usual care.

Study Design & Subject Recruitment: All patients admitted to the pulmonary ward for an AECOPD, will be offered participation into the study. Patients found to have an acute cardiac injury during admission, mobility issues or residence outside the greater Edmonton area will be excluded. Consenting patients will be subsequently randomized into one of three groups: early PR versus late PR versus usual care. Patients randomized to PR will be enrolled within 1 (Early PR; EPR) or 3 months (Late PR; LPR) of discharge into a PR program. Usual care patients will be followed-up by their most responsible physician as determined by the admitting team. The PR group will be enrolled in the Breathe Easy Program at the Center for Lung Health, and will proceed through the program in a typical fashion. All patients will be followed up 6 months after discharge and will be interviewed to assess disease status, management review and if there has been a history of recurrence or relapse of the AECOPD. Hospital admissions and length of stay data will be obtained through electronic medical records. Patient assessments will include: quality of life, 6min walk, dyspnea, self-efficacy, physical activity, pulse wave velocity, vascular function, systemic inflammation (TNFα, MMP-2, IL-6 and CRP) and FeNO. All data will be collected before, immediately after and 6 months after PR. The control group will have the same data collected at the same scheduled time. See above for descriptions of methods.

Data Handling: Data will be entered onto a secure anonymized database.

Data Analysis: The influence of PR on QoL, 6min walk, dyspnea, self-efficacy, physical activity, pulse wave velocity, vascular function, systemic inflammation and eNO will be analyzed using a multivariate mixed-model MANOVA with treatment (Early-PR vs. Late-PR vs. usual care) being a fixed between-group variable and time (pre, immediate post, 6months post) as a repeated variable.

Sample size: Based on previous work, a sample size of 50 in each group (150 total) will be sufficient to detect a between-group differences in QoL, 6min walk, PWV, dyspnea and hospital readmission rates following PR (α=0.05, β=0.8). Based on the investigators recent work, this sample could detect a 10% difference in physical activity following PR (α=0.05, β=0.8). One hundred fifty patients will also allow for stratification of physiological and psychological responses with PR.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the pulmonary ward for an AECOPD will be offered participation into this arm of the study.

Exclusion Criteria:

* Acute cardiac injury during admission
* Mobility issues
* Residence outside the greater Edmonton area

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life - 1 | Change from Baseline Quality of Life - 1 at 8 weeks and 6 months
  Quality of Life - 1 will be assessed using the COPD Assessment tool.
Change in Vascular Function | Change from Baseline Vascular Function at 8 weeks and 6 months
  Vascular function will be assessed using peripheral arterial tone (PAT)
Change in Central and Peripheral Arterial Stiffness (AS) | Change from Baseline Central and Peripheral Arterial Stiffness (AS) at 8 weeks and 6 months
  Arterial Stiffness will be assessed using pulse wave velocity measured from the carotid and femoral (central) and carotid and radial (peripheral) arteries.
Change in Quality of Life - 2 | Change from Baseline Quality of Life - 2 at 8 weeks and 6 months
  Quality of Life - 2 will be assessed using the St. George Respiratory Questionnaire.
Change in Quality of Life - 3 | Change from Baseline Quality of Life - 3 at 8 weeks and 6 months
  Quality of Life - 3 will be assessed using the COPD Self Efficacy Scale.

SECONDARY OUTCOMES:
Change in Inflammatory marker (IL-6) | Change from Baseline IL-6 at 8 weeks and 6 months
  IL-6: is an interleukin that acts as both a pro-inflammatory and anti-inflammatory cytokine.
Change in Inflammatory marker (TNF-alpha) | Change from Baseline TNF-alpha at 8 weeks and 6 months
  TNF-alpha
Change in Inflammatory Marker (MMP-2) | Change from Baseline MMP-2 at 8 weeks and 6 months
  MMP-2
Change in Inflammatory markers (CRP) | Change from Baseline CRP at 8 weeks and 6 months
  CRP: C-reactive protein is a non-specific serum marker of inflammation (range <8 is normal)
Change in Dyspnea (breathlessness) | Change from Baseline Dyspnea at 8 weeks and 6 months
  Dyspnea (breathlessness) will be assessed using Modified Medical Research Council Dyspnea Scale (MMRC)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Stickland, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada